CLINICAL TRIAL: NCT04702802
Title: Clinical Study to Evaluate the Safety of the Viscoelastic Substance PRO-149 When Used as a Device During Phacoemulsification and Intraocular Lens Implantation in Patients With Age-related Cataract, Compared to Healon® EndoCoat.
Brief Title: Study to Evaluate the Safety of the Viscoelastic Substance PRO-149, Compared to Healon® EndoCoat.
Acronym: PRO-149
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOPH149-0220/I
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Age-related Cataract; Phacoemulsification

STUDY DESIGN:
Intervention Model Description: Pilot, controlled, open, comparative, randomized clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1; PRO-149 (Experimental): Viscoelastic substance PRO-149 (sodium hyaluronate 3%) in pre-filled syringe to be applied in the ocular anterior chamber during phacoemulsification surgery in an amount sufficient to form the desired intraocular space and allow the technical maneuvers required for the procedure.
  Interventions: Device: Sodium hyaluronate 3%
- Arm 2; Healon® EndoCoat (Active Comparator): Viscoelastic substance Healon® EndoCoat (sodium hyaluronate 3%) in pre-filled syringe to be applied in the ocular anterior chamber during phacoemulsification surgery in an amount sufficient to form the desired intraocular space and allow the technical maneuvers required for the procedure.
  Interventions: Device: Sodium hyaluronate 3%

INTERVENTIONS:
Device: Sodium hyaluronate 3% — During intraocular surgery phacoemulsification and intraocular lens implantation, patients with age-related cataract will be exposed to injection of viscoelastic device in the anterior chamber, allowing the procedure to take place.
  Other Names: PRO-149
  Arms: Arm 1; PRO-149
Device: Sodium hyaluronate 3% — During intraocular surgery phacoemulsification and intraocular lens implantation, patients with age-related cataract will be exposed to injection of viscoelastic device in the anterior chamber, allowing the procedure to take place.
  Other Names: Healon® EndoCoat
  Arms: Arm 2; Healon® EndoCoat

SUMMARY:
Pilot, controlled, parallel group, open, randomized clinical trial to evaluate the safety of the viscoelastic substance PRO-149 (sodium hyaluronate 3%) after trans-surgical administration as a device in performing phacoemulsification and intraocular lens implantation in 36 patients with age-related cataract, compared to Healon® EndoCoat (sodium hyaluronate 3%).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 49 years old
* Age-related cataract diagnosis which requires phacoemulsification and monofocal intraocular lens implantation
* Being capable of voluntarily grant a signed informed consent.
* Being willing and able to meet the requirements of the study such as attending programmed visits, treatment plan and other study procedures.
* Willingness to be subjected to phacoemulsification and monofocal intraocular lens implantation.
* An anterior chamber depth of ≥ 2.8 mm measured through IOL Master®.
* Pre-surgical cardiologic evaluation that validates the patient's eligibility to surgical procedure, including supporting studies: blood biometry, blood chemistry, clotting time, and electrocardiogram. This evaluation must not exceed 45 days prior to the date of signing of the informed consent.

Exclusion Criteria:

* Previous history of any systemic medical affliction that prevents a patient from being considered eligible for the surgical procedure under sedation and topical anesthesia.
* Previous history of Diabetes Mellitus with A1C ≥ 6.5% (48 mmol/mol) or glucose levels (after no caloric ingestion for ≥ 8 hours) of ≥ 126 mg/dL (7.0 mmol/L).
* Poorly controlled systemic arterial hypertension, defined as a value ≥ 140/90 despite the use of three antihypertensive drugs (one of them a diuretic) at maximum dose.
* Previous history of ocular diseases that may limit the BCVA, or that may reactivate or worsen due to the surgical procedure or due to the use of topical steroids (por example, retinal detachment, macular degeneration, degenerative myopia, proliferative diabetic retinopathy, diabetic macular edema, optic neuritis, uveitis or any other kind of ocular inflammation, glaucoma, intraocular hypertension, corneal dystrophies or ectasias, history of ocular herpes or zoster).
* Active ocular infection
* Pseudoexfoliation syndrome in the eye to withstand surgery, or any other such zonular compromise.
* Pharmacological mydriasis < 6 mm.
* Any congenital anomalies in the eye to withstand surgery.
* Any alteration that prevents a reliable Goldmann tonometry in the eye to withstand surgery.
* IOP >21mmHg in the eye to withstand surgery, or previous history of IOP > 21 mmHg after topical steroid use.
* Corneal endothelial cell count < 1500 cells/mm2 in the eye to withstand surgery.
* Previous history of corneal or intraocular surgery.
* Planned multiple procedures during cataract surgery (for example, trabeculectomy, keratotomies, etc)
* Previous history of ocular trauma in the eye to withstand surgery (including surgical procedures)
* Having one functional eye.
* Having participated in clinical trials within 30 days prior to signing this study's informed consent form.
* Having participated previously in this study.
* Previous history of drug addiction within the last 2 years prior to signing this study's informed consent form.
* Having a previous history of any ophthalmological surgical procedure, within the last 3 months prior to the informed consent signing date.
* Having any kind of programed surgery during the period of this study.
* Being or having any immediate family members (spouse, parent/legal tutor, sibling or child) who work either in the investigation center or for the sponsor of this study.

Min Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Olvera Montaño, MD, Study Director — Regional Medical Affairs Director
Locations (1):
- SalaUno Salud, S.A.P.I. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palacio-Pastrana C, Munoz-Villegas P, Daniel-Dorantes F, Sanchez-Rios A, Olvera-Montano O, Martinez-Montoya YI, Quintana-Hau JD, Baiza-Duran LM. Evaluation of the Rheological Properties, Preclinical Safety, and Clinical Effectiveness of a New Dispersive Ophthalmic Viscoelastic Device for Cataract Surgery. Med Devices (Auckl). 2022 Aug 24;15:293-305. doi: 10.2147/MDER.S379050. eCollection 2022. PMID 36046598

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Cases (Eyes)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat | Total
Number analyzed (Participants) | 18 | 18 | 36
Number analyzed (Cases (Eyes)) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.11 (10.8) | 72.50 (8.8) | 69.89 (15.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 18 | 18 | 36
Corneal Endothelial Cell Count [Mean (Standard Deviation); unit: cells/mm2] — By means of specular microscopy, endothelial cell was performed. Density expressed in cells/mm2 will was recorded. Normal density varies according to age, but an average of 1500 - 3500 cells/mm2 (age 40 to 90) has been described.
  cells/mm2 | 2584.39 (385.5) | 2558.33 (363.4) | 2571.36 (369.45)

OUTCOME MEASURES:

1. Primary Outcome: Change in Corneal Endothelial Cell Count
Description: By means of specular microscopy, endothelial cell count will take place. Density expressed in cells/mm2 will be recorded. Normal density varies according to age, but an average of 1500 - 3500 cells/mm2 (age 40 to 90) has been described.
Time Frame: Days: -15 (±2) (eligibility visit), and 29 (±2) (final visit)
Measure: Mean (Standard Deviation); unit: cells/mm2
Units Other Than Participants: Cases (eyes)
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
Number analyzed (Cases (eyes)) | 18 | 18
cells/mm2 | -441.33 (420.4) | -482.3 (487.7)

2. Primary Outcome: Change in Intraocular Pressure (IOP)
Description: Measured through Goldman tonometer in milligrams of mercury (mmHg). After instillation of topical anesthetic (tetracaine 0.5%) and fluorescein stain, IOP is evaluated twice to obtain an average to be recorded. Normal values are considered between 10 and 21 mmHg.
Time Frame: Days: -15 (±2) (eligibility visit [EV]), 1 (first safety evaluation visit [V1]), 8 (±2) (second safety evaluation visit [V2]), and 29 (±2) (final visit [FV])
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Cases (eyes)
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
Number analyzed (Cases (eyes)) | 18 | 18
mmHg
  EV IOP | 15.83 (2.4) | 15.78 (2.2)
  V1 IOP | 19.28 (7.1) | 16.50 (4.6)
  V2 IOP | 15.78 (2.7) | 15.56 (3.1)
  FV IOP | 15.22 (3.0) | 14.94 (2.7)

3. Secondary Outcome: Number of Participants Presenting Adverse Events
Description: Presence/absence adverse events, defined as the appearance of any unfavorable reaction in a patient participating in a clinical investigation in which any pharmaceutical product is being administered, regardless of the causal attribution.
Time Frame: From Day -15 (±2) (eligibility visit) through Day 29 (±2) (final visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
Participants | 1 | 2

4. Secondary Outcome: Change in Central Corneal Thickness
Description: By means of specular microscopy, corneal thickness will be evaluated, reported in μm.
Time Frame: Days: -15 (±2) (eligibility visit [EV]), and 29 (±2) (final visit [FV])
Measure: Mean (Standard Deviation); unit: μm
Units Other Than Participants: Cases (eyes)
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
Number analyzed (Cases (eyes)) | 18 | 18
μm
  EV Central Corneal Thickness | 517.61 (34.8) | 525.17 (31.5)
  FV Central Corneal Thickness | 527.50 (44.4) | 527.94 (27.6)

5. Secondary Outcome: Change in Anterior Chamber Cellularity
Description: During evaluation with a slit lamp, setting the beam of light to 0.2 mm x 0.2 mm dimensions, it will be obliquely aimed to the anterior chamber. The Standardization of Uveitis Nomenclature (SUN) system was used for grading this variable, according to number of observed cells: grade 0 (none), grade ½+ (1-5 cells), grade 1+ (6-15 cells), grade 2+ (16-25 cells), grade 3+ (26-60 cells), grade 4+ (>60 cells). A higher score represents a worse outcome.
Time Frame: as for outcome 2
Measure: Number; unit: Cases (eyes)
Units Other Than Participants: Cases (eyes)
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
Number analyzed (Cases (eyes)) | 18 | 18
Cases (eyes)
  EV Anterior chamber cellularity : 0 (none) | 18 | 18
  EV Anterior chamber cellularity : 1/2 (1-5) | 0 | 0
  EV Anterior chamber cellularity : 1 + (6-15) | 0 | 0
  EV Anterior chamber cellularity : 2 + (16-25 | 0 | 0
  V1 Anterior chamber cellularity : 0 (none) | 1 | 0
  V1 Anterior chamber cellularity : 1/2 (1-5) | 7 | 5
  V1 Anterior chamber cellularity : 1 + (6-15) | 8 | 9
  V1 Anterior chamber cellularity : 2 + (16-25 | 2 | 4
  V2 Anterior chamber cellularity : 0 (none) | 9 | 9
  V2 Anterior chamber cellularity : 1/2 (1-5) | 8 | 7
  V2 Anterior chamber cellularity : 1 + (6-15) | 1 | 2
  V2 Anterior chamber cellularity : 2 + (16-25 | 0 | 0
  FV Anterior chamber cellularity : 0 (none) | 18 | 18
  FV Anterior chamber cellularity : 1/2 (1-5) | 0 | 0
  FV Anterior chamber cellularity : 1 + (6-15) | 0 | 0
  FV Anterior chamber cellularity : 2 + (16-25 | 0 | 0

6. Secondary Outcome: Change in Anterior Chamber Flare
Description: During evaluation with a slit lamp, setting the beam of light to 0.2 mm x 0.2 mm dimensions, it will be obliquely aimed to the anterior chamber. The Standardization of Uveitis Nomenclature (SUN) system was used for grading this variable: grade 0 (No flare), grade 1+ (Mild), grade 2+ (Moderate; iris and lens clearly visible), grade 3+ (Marked; slightly blurry iris and lens), grade 4+ (>60 cells; fibrin). A higher score represents a worse outcome.
Time Frame: as for outcome 2
Measure: Number; unit: Cases (eyes)
Units Other Than Participants: Cases (eyes)
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
Number analyzed (Cases (eyes)) | 18 | 18
Cases (eyes)
  EV Anterior Chamber Flare : 0 (No flare) | 18 | 18
  EV Anterior Chamber Flare : 1+ (Mild) | 0 | 0
  EV Anterior Chamber Flare : 2+ (Moderate; iris and lens clearly visible) | 0 | 0
  V1 Anterior Chamber Flare : 0 (No flare) | 11 | 6
  V1 Anterior Chamber Flare : 1+ (Mild) | 6 | 11
  V1 Anterior Chamber Flare : 2+ (Moderate; iris and lens clearly visible) | 1 | 1
  V2 Anterior Chamber Flare : 0 (No flare) | 18 | 17
  V2 Anterior Chamber Flare : 1+ (Mild) | 0 | 1
  V2 Anterior Chamber Flare : 2+ (Moderate; iris and lens clearly visible) | 0 | 0
  FV Anterior Chamber Flare : 0 (No flare) | 18 | 18
  FV Anterior Chamber Flare : 1+ (Mild) | 0 | 0
  FV Anterior Chamber Flare : 2+ (Moderate; iris and lens clearly visible) | 0 | 0

7. Secondary Outcome: Change in Best Corrected Visual Acuity (BCVA)
Description: With the patient's best possible refractive correction, visual acuity will be evaluated through the Snellen chart. Its notation (fraction or decimal) is described as the distance from the chart at which the test is performed, divided by the distance at which a letter equals vertically 5 minutes of arc.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: decimal score (Snellen Chart)
Units Other Than Participants: Cases (eyes)
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
Number analyzed (Cases (eyes)) | 18 | 18
decimal score (Snellen Chart)
  EV BCVA | 0.33 (0.19) | 0.42 (0.17)
  V1 BCVA | 0.49 (0.21) | 0.56 (0.24)
  V2 BCVA | 0.81 (0.21) | 0.80 (0.16)
  FV BCVA | 0.93 (0.14) | 0.91 (0.13)

8. Other Pre Specified Outcome: Trans-surgical Evaluation
Description: During the phacoemulsification and intraocular lens implantation, the surgeon will evaluate the performance of the viscoelastic substance used during the procedure trough a questionnaire that will inquire on the following: Capability to maintain a formed anterior chamber during continuous circular capsulorhexis and intraocular lens implantation, retention during phacoemulsification, user-friendliness, ergonomics, ease of use during capsulorhexis, transparency during surgery and ease of use during extraction. Scale: 0 (very bad), 1 (bad), 2 (acceptable), 3 (good), 4 (very good).
Time Frame: Days: 0 (surgery)
Population: (the average performance score across devices)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
Number analyzed (Participants) | 18 | 18
score on a scale | 3.47 (0.6) | 3.50 (0.6)

ADVERSE EVENTS:
Time Frame: From day 1 (basal visit) to the final visit on day 29 (±2 days)
Arm/Group | Arm 1; PRO-149 | Arm 2; Healon® EndoCoat
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1; PRO-149 (N=18) | Arm 2; Healon® EndoCoat (N=18)
conjunctival hyperemia (Eye disorders) | 0 | 1
intraocular hypertension (Eye disorders) | 1 | 0
rupture of the posterior capsule (Eye disorders) | 1 | 0
striations in the descemet membran (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT04702802/Prot_SAP_000.pdf